CLINICAL TRIAL: NCT06926400
Title: A Prospective, Multicenter, Randomized Controlled Clinical Trial to Evaluate the Effectiveness and Safety of the Coronary Artery Serrated Cutting Balloon Dilation Catheter for the Predilation of Coronary Artery Stenosis Lesions
Brief Title: The Effectiveness and Safety of the Coronary Artery Serrated Cutting Balloon Dilation Catheter in the Pre-dilation of Coronary Artery Stenosis Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JW Medical Systems Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JW-SEBC202412
Record Dates: First submitted 2025-04-01; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coronary Artery Serrated Cutting Balloon Dilatation Catheter (Shandong JW Medical Products Co., Ltd. (Experimental)
  Interventions: Device: Coronary artery sawtooth cutting balloon dilation catheter
- Cutting Balloon Catheter (Active Comparator)
  Interventions: Device: Cutting balloon catheter

INTERVENTIONS:
Device: Coronary artery sawtooth cutting balloon dilation catheter — Ninety-one subjects who met the inclusion criteria were enrolled and randomly assigned to the treatment group using a coronary artery sawtooth cutting balloon dilation catheter.
  Arms: Coronary Artery Serrated Cutting Balloon Dilatation Catheter (Shandong JW Medical Products Co., Ltd.
Device: Cutting balloon catheter — Ninety-one subjects who met the inclusion criteria were enrolled and randomly assigned to the treatment group using a cutting balloon catheter.
  Arms: Cutting Balloon Catheter

SUMMARY:
To evaluate the effectiveness and safety of the coronary serrated cutting balloon dilation catheter for the pre-dilation of coronary artery stenosis lesions.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized controlled, non-inferiority designed clinical trial. It is planned to enroll a total of 182 eligible subjects from multiple research centers. The subjects will be randomly assigned to the experimental group (n = 91) and the control group (n = 91) in a 1:1 ratio. All subjects will undergo immediate coronary angiography after percutaneous transluminal coronary angioplasty (PTCA) to evaluate the success rate of the device.

ELIGIBILITY:
Inclusion Criteria:

* ① The age is between 18 and 80 years old (including the boundary values), and the subjects are male or non-pregnant female.

  * Have single or multiple coronary artery lesions and diagnosed ischemic heart disease (for example: stable angina pectoris, unstable angina pectoris, old myocardial infarction or asymptomatic myocardial ischemia).

    * There are coronary artery stenosis lesions confirmed by coronary angiography, which are suitable for percutaneous coronary intervention. The coronary artery stenosis is ≥ 70% (by visual estimation); or ≥ 50% (by visual estimation) and accompanied by evidence of ischemia, and the TIMI blood flow is ≥ Grade 1.

      * There are de novo or restenosis lesions in the coronary arteries of autologous or bypass graft vessels, and interventional treatment is required.

        * The visually estimated reference vessel diameter of the target lesion is 2.0mm - 4.0mm, and the lesion length is ≤ 20mm.

          * When there are multiple lesions that need to be treated, only one coronary artery lesion is selected as the target lesion, and the non-target lesions must be located on different vascular branches.

Be able to understand the purpose of the study, voluntarily participate and sign the informed consent form, and be able to and willing to accept the follow-up as specified in this trial.

Exclusion Criteria:

* General Exclusion Criteria

  * Patients with New York Heart Association (NYHA) Class IV heart failure.

    * Patients with contraindications to anti - platelet and anticoagulant therapy and are unable to receive anticoagulant treatment.

      * Patients who have had any myocardial infarction within one week.

        * Patients with an allergic reaction to contrast agents. ⑤ Patients with severe renal failure, with a serum creatinine level > 2.0 mg/dl (177 μmol/L).

          * Patients who have undergone heart transplantation.

            * Patients who have had active peptic ulcer or active gastrointestinal bleeding within 1 month before surgery.

              ⑧ Patients who have had a stroke or transient ischemic attack within 3 months before surgery.
              * Pregnant or lactating patients. ⑩ Patients who are currently participating in any other clinical trials. ⑪ Patients whom the investigator deems unsuitable for enrollment. Exclusion Criteria Related to the Target Lesion (Detected by Coronary Angiography)
  * Tortuous lesions or lesions with an angulation of ≥ 45 degrees at the lesion site.

    * Lesions at the ostium with a distance of ≤ 2 mm from the left main coronary artery.

      * Unprotected left main coronary artery lesions. ④ Coronary angiography shows the presence of thrombus. ⑤ Before using the test device or the control device, the target lesion has a dissection of Type C or higher.

Target lesions that require treatment with coronary atherectomy or special balloons (such as scored balloons, spiked balloons, shock - wave lithotripsy systems, and cutting balloons of other brands).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Device Procedural Success Rate | one hour

SECONDARY OUTCOMES:
Clinical treatment success rate | one hour
acute lumen gain,ALG | one hour
  Immediate lumen gain is defined as: ALG = the immediate minimum lumen diameter after balloon dilation - the minimum lumen diameter before the operation.
The incidence of the composite endpoint of target lesion failure (TLF) within 30 days after surgery | 30 days
The incidence of patient-related cardiovascular clinical composite endpoint (POCE) within 30 days after surgery | 30 days
The incidence of major adverse cardiac events (MACE) within 30 days after surgery | 30 days
Evaluation of Device Performance | one hour
  CRF
The incidence rate of medical device-related complications | one hour
The incidence rate of device defects | one hour
The incidence rate of adverse events and serious adverse events | thirty days

CONTACTS AND LOCATIONS:
Overall Officials: Yu Bo, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University

IPD SHARING:
Plan to Share IPD: No